CLINICAL TRIAL: NCT03464409
Title: Supporting Patient Decisions About Upper Extremity Surgery in Cervical Spinal Cord Injury (Aim 2)
Brief Title: Supporting Patient Decisions About UE Surgery in Cervical SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); VA St. Louis Health Care System (U.S. Federal Agency); VA Palo Alto Health Care System (U.S. Federal Agency); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201706092
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Cervical Spinal Cord Injury
Keywords: Nerve Transfer Surgery; Tendon Transfer Surgery; Decision Support Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SCI Patient - Nerve Transfer Surgery (Active Comparator): Patients aged 18 to 80 with a mid cervical level spinal cord injury seeking nerve transfer surgery to improve hand and arm function. Participants will be assessed at 3 time points: Baseline (pre-operatively), Early Followup (1 month post-operatively) and Late Followup (6-24 months later). Assessments will include the Spinal Cord Independence Measure (SCIM-SR), the 36-Item Short Form Health Survey (SF-36), and a semi-structured interview to be conducted by a study team member.
  Interventions: Other: Semi-structured interview; Other: Spinal Cord Independence Measure (SCIM-SR); Other: SF-36
- SCI Patient - Tendon Transfer Surgery (Active Comparator): Patients aged 18 to 80 with a mid cervical level spinal cord injury seeking tendon transfer surgery to improve hand and arm function. Participants will be assessed at 3 time points: Baseline (pre-operatively), Early Followup (1 month post-operatively) and Late Followup (6-24 months later). Assessments will include the Spinal Cord Independence Measure (SCIM-SR), the 36-Item Short Form Health Survey (SF-36), and a semi-structured interview to be conducted by a study team member.
  Interventions: Other: Semi-structured interview; Other: Spinal Cord Independence Measure (SCIM-SR); Other: SF-36
- SCI Patient - No Surgery (Active Comparator): Patients aged 18 to 80 with a mid cervical level spinal cord injury who did not chose to have surgery to improve hand and arm function. Participants will be assessed at 3 time points: Baseline, Early Followup (1 month later), and Late Followup (6-24 months later). Assessments will include the Spinal Cord Independence Measure (SCIM-SR), the 36-Item Short Form Health Survey (SF-36), and a semi-structured interview to be conducted by a study team member.
  Interventions: Other: Semi-structured interview; Other: Spinal Cord Independence Measure (SCIM-SR); Other: SF-36

INTERVENTIONS:
Other: Semi-structured interview — Semi-structured interviews to be conducted by a study team member.
Other: Spinal Cord Independence Measure (SCIM-SR) — The Spinal Cord Independence Measure - Self Report (SCIM-SR) is a self-report instrument for assessing functional independence of persons with spinal cord injury.
Other: SF-36 — A health-related quality of life (QoL) self-reported survey.

SUMMARY:
The goal of this study is to collect and describe patient and caregiver reported outcomes regarding surgical and non-surgical treatment for improving hand and arm function in the setting of cervical spinal cord injury. Eligible study participants will be recruited across the 4 sites and the investigators plan to recruit the following groups and numbers of participants:

1. Nerve or tendon transfer recipients: people who have elected to undergo nerve (N=10) or tendon (N=10) transfer surgery to restore some hand and arm function as part of their standard clinical care and their caregiver (N=20)
2. Non-surgical control group: people with cervical SCI (N=20) and their caregiver (N=20)

DETAILED DESCRIPTION:
At present, there is limited information that provides the exact time course and probability of gain in specific function (such as hand function) that might help patients and clinicians make decisions regarding novel and time-sensitive surgical treatment options.

Understanding the pros and cons of any surgical intervention, especially in the setting of complex and often incomplete information, is challenging. Ultimately, this project will create a decision support intervention (DSI) that can be used to help clinicians and people living with cervical level SCI and their caregivers. It will be most useful to those with acute or sub-acute injury (< 1year after SCI) for both military personnel and the general public. Clinicians and patients will have evidence to help them make decisions about treatments to improve upper extremity function.

In such a manner, patients can make more well-informed choices that are consistent with their values, needs and goals.

ELIGIBILITY:
CERVICAL SPINAL CORD INJURY PARTICIPANTS

Inclusion criteria:

* Adult subjects (≥18 years and < 80 years) with cervical level SCI ASIA A, B or C (minimum 6 months and maximum 20 years post-injury).

Exclusion criteria:

* Patient who chooses simultaneous tendon and nerve transfer procedure (this would preclude separation of the influence of one surgery compared to the other)
* Patient has ASIA D status (these patients may have progressive return of functionally useful motor function below the level of the SCI and would not routinely be offered acute surgical intervention and their experiences are less-relevant to the target patient population).

CAREGIVER PARTICIPANTS

Inclusion criteria:

* At least 18 years of age
* Able to answer questions about the primary participant's experiences with cervical spinal cord injury

Exclusion criteria:

* The caregiver/spouse declines to participate in the study. Note: Caregiver participation is preferred, but not required, for SCI participant enrollment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Qualitative (interview) Analysis | 24 months
  All interviews will be transcribed verbatim and analyzed using standard qualitative text analysis. Members of the research team will read the transcripts for accuracy and to determine potential topics for coding. The investigators will develop a codebook using inductive and deductive codes. Deductive codes will be directly linked to our research questions. Adding inductive codes, where topics and codes are not pre-determined but are derived directly from the data, will allow the research team to develop a sense of how patients experience the surgical process, and allows for unexpected findings to emerge. Once the codebook is determined, two members of the research team will code the transcripts. Codes will be compared between raters. The investigators will use the codes to infer themes in the data.

SECONDARY OUTCOMES:
Quantitative (survey) Data Analysis | 24 months
  The data analysis will be conducted within each group. To account for correlations among repeated measures from the same patient, the longitudinal data will be analyzed using a mixed model to examine the change in survey outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Ida K Fox, MD, Principal Investigator — Washington University School of Medicine
Locations (4):
- United States (4):
  - Veterans Affairs Palo Alto Health Care System, Palo Alto, California
  - Stanford University, Stanford, California
  - Veterans Affairs St. Louis Health Care System, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fox IK, Davidge KM, Novak CB, Hoben G, Kahn LC, Juknis N, Ruvinskaya R, Mackinnon SE. Nerve Transfers to Restore Upper Extremity Function in Cervical Spinal Cord Injury: Update and Preliminary Outcomes. Plast Reconstr Surg. 2015 Oct;136(4):780-792. doi: 10.1097/PRS.0000000000001641. PMID 26397252
- [Background] Fox IK, Davidge KM, Novak CB, Hoben G, Kahn LC, Juknis N, Ruvinskaya R, Mackinnon SE. Use of peripheral nerve transfers in tetraplegia: evaluation of feasibility and morbidity. Hand (N Y). 2015 Mar;10(1):60-7. doi: 10.1007/s11552-014-9677-z. PMID 25767422
- [Background] Curtin CM, Gater DR, Chung KC. Upper extremity reconstruction in the tetraplegic population, a national epidemiologic study. J Hand Surg Am. 2005 Jan;30(1):94-9. doi: 10.1016/j.jhsa.2004.10.007. PMID 15680562
- [Background] Bertelli JA, Ghizoni MF, Tacca CP. Transfer of the teres minor motor branch for triceps reinnervation in tetraplegia. J Neurosurg. 2011 May;114(5):1457-60. doi: 10.3171/2010.12.JNS101519. Epub 2011 Jan 21. PMID 21250798
- [Background] Bertelli JA, Ghizoni MF. Nerve transfers for elbow and finger extension reconstruction in midcervical spinal cord injuries. J Neurosurg. 2015 Jan;122(1):121-7. doi: 10.3171/2014.8.JNS14277. PMID 25343189
- [Background] Bertelli JA, Tacca CP, Ghizoni MF, Kechele PR, Santos MA. Transfer of supinator motor branches to the posterior interosseous nerve to reconstruct thumb and finger extension in tetraplegia: case report. J Hand Surg Am. 2010 Oct;35(10):1647-51. doi: 10.1016/j.jhsa.2010.07.012. PMID 20888500
- [Background] Friden J, Gohritz A. Brachialis-to-extensor carpi radialis longus selective nerve transfer to restore wrist extension in tetraplegia: case report. J Hand Surg Am. 2012 Aug;37(8):1606-8. doi: 10.1016/j.jhsa.2012.05.005. Epub 2012 Jun 30. PMID 22749482
- [Background] Curtin CM, Hayward RA, Kim HM, Gater DR, Chung KC. Physician perceptions of upper extremity reconstruction for the person with tetraplegia. J Hand Surg Am. 2005 Jan;30(1):87-93. doi: 10.1016/j.jhsa.2004.08.014. PMID 15680561
- [Background] Wagner JP, Curtin CM, Gater DR, Chung KC. Perceptions of people with tetraplegia regarding surgery to improve upper-extremity function. J Hand Surg Am. 2007 Apr;32(4):483-90. doi: 10.1016/j.jhsa.2007.01.015. PMID 17398358
- [Background] Fox PM, Suarez P, Hentz VR, Curtin CM. Access to surgical upper extremity care for people with tetraplegia: an international perspective. Spinal Cord. 2015 Apr;53(4):302-5. doi: 10.1038/sc.2015.3. Epub 2015 Feb 17. PMID 25687516
- [Background] Anderson KD, Friden J, Lieber RL. Acceptable benefits and risks associated with surgically improving arm function in individuals living with cervical spinal cord injury. Spinal Cord. 2009 Apr;47(4):334-8. doi: 10.1038/sc.2008.148. Epub 2008 Nov 25. PMID 19030014
- [Background] Cain SA, Gohritz A, Friden J, van Zyl N. Review of Upper Extremity Nerve Transfer in Cervical Spinal Cord Injury. J Brachial Plex Peripher Nerve Inj. 2015 Aug 6;10(1):e34-e42. doi: 10.1055/s-0035-1558427. eCollection 2015 Dec. PMID 27917237
- [Background] Joseph-Williams N, Newcombe R, Politi M, Durand MA, Sivell S, Stacey D, O'Connor A, Volk RJ, Edwards A, Bennett C, Pignone M, Thomson R, Elwyn G. Toward Minimum Standards for Certifying Patient Decision Aids: A Modified Delphi Consensus Process. Med Decis Making. 2014 Aug;34(6):699-710. doi: 10.1177/0272989X13501721. Epub 2013 Aug 20. PMID 23963501
- [Background] Stacey D, Legare F, Col NF, Bennett CL, Barry MJ, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L, Wu JH. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2014 Jan 28;(1):CD001431. doi: 10.1002/14651858.CD001431.pub4. PMID 24470076
- See also: Center for Nerve Injury & Paralysis, Washington University in St. Louis School of Medicine — http://nerve.wustl.edu